CLINICAL TRIAL: NCT02729220
Title: Respiratory and Cardiovascular Effects in COPD - Report From a Bronchoscopy Investigation Based on the Obstructive Lung Disease In the Northern Sweden (OLIN) Studies
Brief Title: Respiratory and Cardiovascular Effects in COPD
Acronym: KOLIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Annelie F Behndig, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Dr Annelie F Behndig, MD PhD, Investigator, University Hospital, Umeå
Organization: University Hospital, Umeå (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-147_31M
Record Dates: First submitted 2016-02-24; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Aging; Oxidative stress; Proteases; Bronchoscopy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy controls (Other): Bronchoscopy with collection of bronchial biopsies and lavages Arterial stiffness
  Interventions: Other: Bronchoscopy
- Smokers (Other): Bronchoscopy with collection of bronchial biopsies and lavages Arterial stiffness
  Interventions: Other: Bronchoscopy
- COPD rapid decline (Other): Bronchoscopy with collection of bronchial biopsies and lavages Arterial stiffness
  Interventions: Other: Bronchoscopy
- COPD slow decline (Other): Bronchoscopy with collection of bronchial biopsies and lavages Arterial stiffness
  Interventions: Other: Bronchoscopy

INTERVENTIONS:
Other: Bronchoscopy — Sampling of airways

SUMMARY:
The purpose of this study is to find out if subjects with chronic obstructive pulmonary disease have signs of accelerated ageing in their airways.

DETAILED DESCRIPTION:
The age-related impairment of innate immunity and antioxidant defenses likely impacts on development and disease progression of chronic obstructive pulmonary disease, COPD. It has been suggested that aging-related declines in function are accelerated in COPD due to recurrent cycles of inflammation, tissue injury and repair, associated with long-term exposure to cigarette smoke or other airway irritants. Here, the investigators aim to follow up on previous observations of impaired antioxidant responses in the lung of COPD patients, to establish the extent to which this reflects an accelerated aging phenotype, to characterize the molecular mechanisms resulting in this functional deficiency. The proposed studies will employ well-characterized patients with COPD of varying severity and smoking habits, as well as carefully age and smoking history-matched controls. Accelerated aging within the COPD lung will be assessed in endobronchial mucosal biopsies and airway macrophages by assessment of established senescence markers using immunohistochemical, biochemical and PCR-based methods. These markers of tissue age will then be related to the functional activation of transcription factors, known to be induced by oxidative stress and related to cytoprotection such as Nrf2 and AP1. The investigators will also examine whether COPD is associated with an enhanced secretion of inflammatory mediators from senescent cells, consistent with the accelerated aging paradigm and establish how this influences cell function. Deficiencies in metal handling, antioxidant defenses and diminished airway innate immune defenses at the air-lung interface will be assessed. The aim is to identify biomarkers for the risk of rapid lung function deterioration in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD, GOLD stage 2-3.
* Smoking history of at least 10 packyears.

Exclusion Criteria:

* Severe ischemic heart disease.
* Other severe disease.
* Respiratory infection within four weeks.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cellular senescence marker - Ki67 | Baseline
  Endobronchial mucosal biopsies collected by bronchoscopy. Immunohistochemistry for the cellular senescence markers Ki67 will be performed.
Matrix metalloproteinase 12 (MMP12) and the inhibitor TIMP1 | Baseline
  Airway lavages collected by bronchoscopy and serum will be analysed for MMP and TIMP using ELISAs.
Levels of oxidized proteins, 4 HNE | Baseline
  The accumulation of oxidized proteins, 4-Hydroxynonenal, will be assessed in bronchial biopsies.
Antioxidant-related transcription factor Nrf2 | Baseline
  Nuclear factor (erythroid-derived 2)-like 2 (Nrf2) is a transcription factor known to be induced by oxidative stress and related to cytoprotection.

SECONDARY OUTCOMES:
Metals in airway lavages | Baseline
  Airway lavages collected by bronchoscopy will be analysed for metals using mass spectrometry
Lymphocyte subsets in bronchoalveolar lavage | Baseline
  Airway lavages collected by bronchoscopy will be analysed for lymphocyte subsets using flow cytometry.
Arterial stiffness | Baseline
  Non-invasive measurement of arterial stiffness

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health and Clinical Medicine, Division of medicine, Pulmonary medicine, Umeå, Sverige, Sweden

REFERENCES:
- [Derived] Eriksson Strom J, Pourazar J, Linder R, Blomberg A, Lindberg A, Bucht A, Behndig AF. Airway regulatory T cells are decreased in COPD with a rapid decline in lung function. Respir Res. 2020 Dec 14;21(1):330. doi: 10.1186/s12931-020-01593-9. PMID 33317530
- [Derived] Eriksson Strom J, Pourazar J, Linder R, Blomberg A, Lindberg A, Bucht A, Behndig AF. Cytotoxic lymphocytes in COPD airways: increased NK cells associated with disease, iNKT and NKT-like cells with current smoking. Respir Res. 2018 Dec 7;19(1):244. doi: 10.1186/s12931-018-0940-7. PMID 30526599